CLINICAL TRIAL: NCT05298384
Title: Pathophysiologic Study to Understand and Possibly Treat Nocturia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed prior to enrollment of participants.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-00542
Record Dates: First submitted 2022-03-18; First posted 2022-03-28 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Stockings, Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Individuals with nocturia as a result of idiopathic edema and autonomic failure will be assigned to wearing knee high then thigh high compression stockings to assess the effect on weight gain during the day and the number of nocturia events.
  Interventions: Other: Compression stockings

INTERVENTIONS:
Other: Compression stockings — Graduated compression stockings (GCS) are used to treat chronic venous diseases and edema. They help to improve blood flow and prevent blood pooling in the legs. The use of GCS will be in accordance with this indication. The greatest pressure is exerted at the ankle with gradually decreasing pressures up the length of the stockings. GCS are designed for use out of bed and are manufactured using strict medical and technical specifications.

SUMMARY:
This study will mainly look at how well compression stockings decrease body weight between morning and night and the number of nocturia events, by preventing blood from pooling in your legs. Also, this research study is being done to collect the thoughts/reactions/opinions on how nocturia affects the life of one who suffers from nocturia.

DETAILED DESCRIPTION:
This study intends to investigate the different causes nocturia. Patients with nocturia will be assigned to wearing knee high then thigh high compression stockings to assess the effect on weight gain during the day and the number of nocturia events. Renin and aldosterone levels will also be assessed. Furthermore, fluorescein dye will be used to to demonstrate vascular leakage of the fluorescent dye.

ELIGIBILITY:
Inclusion Criteria:

* Age above or equal to 18 years at the time of signing informed consent
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study prior to initiation of any protocol-mandated procedures.

Exclusion Criteria:

* Suspected or proven peripheral arterial disease, including history of peripheral arterial bypass grafting
* Any sensory impairment such as severe peripheral neuropathy as evidenced by patient reported intermittent claudication and/or signs of ischemia such as "blue toes".
* Allergy to stocking textile material.
* Leg edema or pulmonary edema from congestive heart failure.
* Local skin or soft-tissue condition, including recent skin graft, gangrene, oozing dermatitis and severe cellulitis.
* Extreme deformity of the leg, or unusual leg shape or size that would prevent correct fit.
* Treatment with any diuretics such as furosemide or hydrochlorothiazide.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in the level of nocturia | Baseline, Day 11-20 visit, Day 21-30 visit
  To measure the reduction of nocturia by the absolute change in body weight between morning and night and nocturia events at baseline and after compression stocking use.
Change in the quality of life for people with nocturia | Baseline visit, Day 20 visit
  To measure the effect of nocturia on Quality of Life by the percent change in QOL score when comparing baseline and 20 days of treatment with compression stockings.

CONTACTS AND LOCATIONS:
Overall Officials: John Maesaka, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to John.Maesaka@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.